CLINICAL TRIAL: NCT06029712
Title: Developing a Heart Failure Polypill to Improve Outcomes at a Safety Net Hospital: A Pilot Crossover Randomized Controlled Trial
Brief Title: Heart Failure Polypill at a Safety Net Hospital
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23-39360
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure With Reduced Ejection Fraction; HIV Infections
Keywords: Medication adherence; Polypill
MeSH Terms: conditions — HIV Infections; Medication Adherence | interventions — Tin Fluorides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- GDMT delivered in a heart failure polypill (Experimental): The polypill intervention will be pharmacy-level over-encapsulation of heart failure medications (beta-blocker, SGLT2 inhibitor, mineralocorticoid receptor antagonist, and ACE/ARB/ARNI) into a single capsule. For patients on twice-daily sacubitril/valsartan, one dose will be included in the polypill and the second dose will be dispensed separately. The investigators will partner with a local community pharmacy with proficiency in over-encapsulation. For patients in the polypill arm, heart failure medications will be filled as usual, but rather than dispensing each medication separately, the pharmacy technician will hand-pack all once-daily heart failure medications into a small vegan capsule.
  Interventions: Drug: Heart failure polypill
- GDMT delivered as individual tablets (Active Comparator): As described above, participants who are not already prescribed a beta blocker, SGLT2i, ACE/ARB/ARNI, and MRA will be initiated on these medications prior to randomization if no contraindications exist. Participants randomized to usual care will receive their heart failure medications as individual pills. They will have the option to receive medications by mail, clinic pick-up, or pharmacy pick-up.
  Interventions: Drug: Control Rx

INTERVENTIONS:
Drug: Heart failure polypill — Copackaging of heart failure medications (beta blocker, SGLT2i, MRA, and ACE/ARB/ARNI) in an overencapsulated polypill. Individual tablets will be hand-packed into a single capsule at the level of the pharmacy. Specific medications and doses will be individualized to the participant.
  Arms: GDMT delivered in a heart failure polypill
Drug: Control Rx — GDMT delivered as individual tablets
  Arms: GDMT delivered as individual tablets

SUMMARY:
A novel four-drug regimen for heart failure with reduced ejection fraction (HFrEF) extends patients' life expectancy by an average of 6 years compared to traditional therapies, in addition to improving quality of life. Unfortunately, uptake of this complex multi-drug regimen has been low, especially among underserved communities with barriers to medication adherence. Although combination tablets have transformed access to care for conditions such as HIV and tuberculosis, no combination pill is available for HFrEF.

In the proposed study, the investigators will utilize inexpensive over-encapsulation techniques to develop a novel combination pill ("polypill") for patients with HFrEF. In Aim 1, the investigators will conduct stakeholder interviews with patients, providers, and pharmacists to inform the design of a HFrEF polypill. In Aim 2, the investigators will conduct a pilot, single-center, crossover randomized clinical trial to investigate whether, compared to usual care, a HFrEF polypill increases medication adherence among 20-40 adults with HFrEF. Given the high daily pill burden among patients with HIV and HFrEF, the investigators aim to recruit a subgroup of patients with HIV (~10-20 participants) in addition to a subgroup of patients without HIV (~10-20 participants).

DETAILED DESCRIPTION:
Hypothesis: Compared with usual care, a HFrEF polypill implementation strategy will increase adherence to GDMT 4 weeks and reduce total daily pill burden among patients with HFrEF.

Rationale:HFrEF among PWH is associated with a high pill burden, which adversely impacts adherence. Over-encapsulation is an inexpensive and replicable method to co-package several tablets into a single capsule at the level of the pharmacy. However, the role of over-encapsulation to reduce pill burden among adults with HIV and HFrEF is unknown.

Design: Pilot phase II open-label randomized trial with a 2x2 crossover design (AB/BA)

Intervention: The intervention will be pharmacy-level over-encapsulation of once-daily heart failure medications (beta-blocker, SGLT2 inhibitor, spironolactone, and ACE/ARB/ARNI) into a single capsule. For some patients, other once-daily cardiovascular medications, such as a diuretic, may be included if capsule size allows (otherwise, these medications will continued to be filled separate to the polypill, as individual tablets). If the patient uses a twice-daily ARNI medication, the morning dose may be included in the polypill and the PM dose will continue to be dispensed separately. The investigators will partner with Daniel's Pharmacy, a local community pharmacy with proficiency in over-encapsulation and over 20 years' experience working with ZSFG to deliver adherence interventions.

Polypill Description: For patients in the polypill arm, heart failure medications will be filled as usual, but rather than dispensing each medication separately, the pharmacy technician will hand-pack all once-daily heart failure medications into a small plastic capsule. The doses will be individualized to the patient based on their physician's prescription. Thus, the polypill will be a late-stage implementation intervention to reduce pill burden, without restricting dose possibilities or interfering with medication titration.

Visit Schedule and Randomization: Patients will first attend an intake visit (week T-1), where eligibility will be reviewed, informed consent will be obtained, baseline patient questionnaires will be collected, and additional GDMT agents may be prescribed by the study clinician if clinically indicated and there are no contraindications. At the first trial visit (week 0), baseline labs will be collected and additional GDMT agents may prescribed if clinically indicated, with the goal of all participants being prescribed guideline-directed quad therapy for HFrEF prior to randomization if there are no contraindications.

During the first trial visit (week 0), half of participants will be randomized to the AB group (polypill for 4 weeks, then individual tablets for 4 weeks). The other half of participants will be randomized to the BA group (individual tablets for 4 weeks, then polypill for 4 weeks).

After randomization, participants assigned to receive the polypill up-front will be delivered 30-day supplies of the polypill via their preferred delivery method (mail, pick up at a ZSFG clinic, or pick up at Daniel's Pharmacy). Participants assigned to usual care will be mailed or pick up their existing heart failure medications as individual pills. The screening visit and first trial visit may be timed by study clinicians based on when the participant's heart failure medications will be ready for a refill according to insurance.

At trial follow-up visits at 4 and 8 weeks, participants will be assessed for outcomes and adverse events and will undergo lab monitoring as clinically indicated. Patients will be asked to bring in their pill bottles and/or MediSets or bubble packs. Medication doses may be titrated at these visits if clinically indicated. Participants in the AB and BA arms will have the same follow-up schedule, and can opt to receive refills of their medications by mail, at the pharmacy, or in clinic. Any new starts of guideline-directed heart failure medications that are included in the polypill will be continued as individual pills when the polypill group crosses over to the individual tablet condition, and/or when the trial concludes. All participants will be referred to cardiology clinic, if not already established there, for ongoing management of their heart failure therapies after the trial.

ELIGIBILITY:
Inclusion criteria:

* Adults age 18+ with heart failure (current or prior NYHA stage II-IV)
* Ejection fraction <50% on the most recent echocardiogram or MRI
* Last eGFR > 30
* Able to conveniently obtain medications through one of 3 available mechanisms (mail, pick up at a ZSFG clinic, or pick up at Daniel's pharmacy)
* Working phone number for telephone visits
* In addition to the inclusion criteria above, the investigators will preferentially recruit the following patient groups: people with HIV for a recruitment subgroup; patients who are less connected to cardiology care; people who are on <4 pillars of GDMT, and have difficulty with medication adherence (as evidenced by detectable HIV viral load or refill gaps in Epic); and people who do not use bubble packs and do not have daily medication support staff for med administration.

Exclusion criteria:

* Patients who are not fluent in English (due to constraints of the small pilot trial)
* Patients who are incarcerated
* Patients who cannot provide informed consent
* Patients with a ventricular assist device (VAD) or patients with an MI, unstable angina, stroke, or TIA within 12 weeks prior to enrollment
* Women who are pregnant, breastfeeding or of childbearing potential and are not using and do not plan to continue using medically acceptable form of contraception throughout the study (pharmacological or barrier methods).
* Concomitant medical condition which in the opinion of the study team could interfere with the safe conduct of the study including outcome assessment.
* Participation in a concurrent interventional medical investigation or pharmacologic clinical trial. Patients in observational, natural history or epidemiological studies not involving an intervention are eligible.
* Participant's responsible physician believes it is not appropriate for participant to take part in the study.
* Unable to complete study procedures and/or plan to move out of the study area in the next 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2025-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colette DeJong, MD, Principal Investigator — University of California, San Francisco; Priscilla Hsue, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Pandey A, Keshvani N, Wang TJ. Should Polypills Be Used for Heart Failure With Reduced Ejection Fraction? Circulation. 2022 Jul 26;146(4):276-278. doi: 10.1161/CIRCULATIONAHA.122.059661. Epub 2022 Jul 25. No abstract available. PMID 35877830
- [Background] Gnanenthiran SR, Agarwal A, Patel A. Frontiers of cardiovascular polypills: From atherosclerosis and beyond. Trends Cardiovasc Med. 2023 Apr;33(3):182-189. doi: 10.1016/j.tcm.2021.12.013. Epub 2021 Dec 30. PMID 34973412
- [Background] Mastromarino V, Casenghi M, Testa M, Gabriele E, Coluccia R, Rubattu S, Volpe M. Polypharmacy in heart failure patients. Curr Heart Fail Rep. 2014 Jun;11(2):212-9. doi: 10.1007/s11897-014-0186-8. PMID 24493574
- [Background] Castellano JM, Pocock SJ, Bhatt DL, Quesada AJ, Owen R, Fernandez-Ortiz A, Sanchez PL, Marin Ortuno F, Vazquez Rodriguez JM, Domingo-Fernandez A, Lozano I, Roncaglioni MC, Baviera M, Foresta A, Ojeda-Fernandez L, Colivicchi F, Di Fusco SA, Doehner W, Meyer A, Schiele F, Ecarnot F, Linhart A, Lubanda JC, Barczi G, Merkely B, Ponikowski P, Kasprzak M, Fernandez Alvira JM, Andres V, Bueno H, Collier T, Van de Werf F, Perel P, Rodriguez-Manero M, Alonso Garcia A, Proietti M, Schoos MM, Simon T, Fernandez Ferro J, Lopez N, Beghi E, Bejot Y, Vivas D, Cordero A, Ibanez B, Fuster V; SECURE Investigators. Polypill Strategy in Secondary Cardiovascular Prevention. N Engl J Med. 2022 Sep 15;387(11):967-977. doi: 10.1056/NEJMoa2208275. Epub 2022 Aug 26. PMID 36018037
- [Background] Mohd Salleh NA, Richardson L, Kerr T, Shoveller J, Montaner J, Kamarulzaman A, Milloy MJ. A Longitudinal Analysis of Daily Pill Burden and Likelihood of Optimal Adherence to Antiretroviral Therapy Among People Living With HIV Who Use Drugs. J Addict Med. 2018 Jul/Aug;12(4):308-314. doi: 10.1097/ADM.0000000000000403. PMID 29521670
- [Background] Baldridge AS, Huffman MD, Lazar D, Abbas H, Flowers FM, Quintana A, Jackson A, Khan SS, Chopra A, Vu M, Tripathi P, Jacobson T, Sanuade OA, Kandula NR, Persell SD, Paparello JJ, Rosul LL, Mejia J, Lloyd-Jones DM, Chow CK, Ciolino JD. Efficacy and safety of a quadruple ultra-low-dose treatment for hypertension (QUARTET USA): Rationale and design for a randomized controlled trial. Am Heart J. 2022 Dec;254:183-193. doi: 10.1016/j.ahj.2022.09.004. Epub 2022 Sep 15. PMID 36116516
- [Background] Chow CK, Thakkar J, Bennett A, Hillis G, Burke M, Usherwood T, Vo K, Rogers K, Atkins E, Webster R, Chou M, Dehbi HM, Salam A, Patel A, Neal B, Peiris D, Krum H, Chalmers J, Nelson M, Reid CM, Woodward M, Hilmer S, Thom S, Rodgers A. Quarter-dose quadruple combination therapy for initial treatment of hypertension: placebo-controlled, crossover, randomised trial and systematic review. Lancet. 2017 Mar 11;389(10073):1035-1042. doi: 10.1016/S0140-6736(17)30260-X. Epub 2017 Feb 10. PMID 28190578
- [Background] Bahiru E, de Cates AN, Farr MR, Jarvis MC, Palla M, Rees K, Ebrahim S, Huffman MD. Fixed-dose combination therapy for the prevention of atherosclerotic cardiovascular diseases. Cochrane Database Syst Rev. 2017 Mar 6;3(3):CD009868. doi: 10.1002/14651858.CD009868.pub3. PMID 28263370
- [Background] Vijay A, Mohanan PP, Kondal D, Baldridge A, Davies D, Devarajan R, Unni G, Abdullakutty J, Natesan S, Joseph J, Jayagopal PB, Joseph S, Gopinath R, Prabhakaran D, Huffman MD, Agarwal A. Polypill Eligibility for Patients with Heart Failure With Reduced Ejection Fraction in South India: A Secondary Analysis of a Prospective, Interrupted Time Series Study. J Am Heart Assoc. 2021 Oct 19;10(20):e021676. doi: 10.1161/JAHA.121.021676. Epub 2021 Oct 6. No abstract available. PMID 34612082
- [Background] Munoz D, Uzoije P, Reynolds C, Miller R, Walkley D, Pappalardo S, Tousey P, Munro H, Gonzales H, Song W, White C, Blot WJ, Wang TJ. Polypill for Cardiovascular Disease Prevention in an Underserved Population. N Engl J Med. 2019 Sep 19;381(12):1114-1123. doi: 10.1056/NEJMoa1815359. PMID 31532959
- [Background] Castellano JM, Sanz G, Penalvo JL, Bansilal S, Fernandez-Ortiz A, Alvarez L, Guzman L, Linares JC, Garcia F, D'Aniello F, Arnaiz JA, Varea S, Martinez F, Lorenzatti A, Imaz I, Sanchez-Gomez LM, Roncaglioni MC, Baviera M, Smith SC Jr, Taubert K, Pocock S, Brotons C, Farkouh ME, Fuster V. A polypill strategy to improve adherence: results from the FOCUS project. J Am Coll Cardiol. 2014 Nov 18-25;64(20):2071-82. doi: 10.1016/j.jacc.2014.08.021. Epub 2014 Sep 1. PMID 25193393
- [Derived] DeJong C, Durstenfeld MS, Davis JD, Wang CS, Riley ED, Huffman MD, Hickey MD, Shade SB, Chen JC, Kazi DS, Grochowski J, Steward WT, Zier LS, Moreau N, Sandhu AT, Heidenreich PA, Agarwal A, Hsue PY. Delivering guideline-directed medical therapy for heart failure with reduced ejection fraction as an over-encapsulated polypill: rationale and protocol for the COMBO-HF-X pilot crossover randomised clinical trial. BMJ Open. 2025 Mar 21;15(3):e093663. doi: 10.1136/bmjopen-2024-093663. PMID 40118491

RESULTS

PARTICIPANT FLOW:
Groups:
- GDMT Delivered in a Heart Failure Polypill First (Individual Tablets Second): The polypill intervention will be pharmacy-level over-encapsulation of heart failure medications (beta-blocker, SGLT2 inhibitor, mineralocorticoid receptor antagonist, and ACE/ARB/ARNI) into a single capsule. For patients on twice-daily sacubitril/valsartan, one dose will be included in the polypill and the second dose will be dispensed separately. The investigators will partner with a local community pharmacy with proficiency in over-encapsulation. For patients in the polypill arm, heart failure medications will be filled as usual, but rather than dispensing each medication separately, the pharmacy technician will hand-pack all once-daily heart failure medications into a small vegan capsule. This group is assigned to polypill first and individual tablets second.
- GDMT Delivered as Individual Tablets First (Polypill Second): As described above, participants who are not already prescribed a beta blocker, SGLT2i, ACE/ARB/ARNI, and MRA will be initiated on these medications prior to randomization if no contraindications exist. Participants randomized to usual care will receive their heart failure medications as individual pills. They will have the option to receive medications by mail, clinic pick-up, or pharmacy pick-up. After 1 month, participants assigned to individual tablets first will be switched to the polypill intervention.
Period: Overall Study
Arm/Group | GDMT Delivered in a Heart Failure Polypill First (Individual Tablets Second) | GDMT Delivered as Individual Tablets First (Polypill Second)
Started | 17 | 18
Completed | 14 | 13
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GDMT Delivered in a Heart Failure Polypill First (Individual Tablets Second) | GDMT Delivered as Individual Tablets First (Polypill Second) | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age in years
  years | 55 [52 to 60] | 50.5 [42 to 61] | 54 [46 to 61]
Sex: Female, Male [Count of Participants; unit: Participants] — Sex
  Participants
    Female | 2 | 7 | 9
    Male | 15 | 11 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Black or African American | 11 | 7 | 18
    White | 3 | 7 | 10
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 2 | 4 | 6
    Not Hispanic or Latino | 15 | 14 | 29
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Measured Adherence to GDMT by Pill Count
Description: The primary outcome will be overall adherence to GDMT, as determined by pill count. We will first calculate the % adherence ratio for each prescribed class of GDMT (# pills missing / # pills supposed to be missing). The adherence ratio for each prescribed class of GDMT will then be averaged to derive the overall adherence ratio to GDMT. Pill count may be performed in-office or over videoconferencing.
Time Frame: The outcome will be measured 1) following a month of polypill use, and 2) following a month of individual tablet use.
Population: As part of the crossover analysis, the individual tablet periods were combined from both assignment groups (individual tablets first and polypill first), and the polypill periods were combined.
Measure: Mean (95% Confidence Interval); unit: adherence ratio expressed in %
Groups:
- Individual Tablets: This group represents the period of time during which participants were assigned to HF GDMT with individual tablets.
- Polypill: This group represents the period of time during which participants were assigned to HF GDMT with a polypill.
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 27 | 27
adherence ratio expressed in % | 74.6 [66.6 to 82.5] | 83.3 [75.3 to 91.3]

2. Secondary Outcome: Morisky Medication Adherence-8 (MMAS-8) Questionnaire
Description: The MMAS-8 scale consists of 8 items. Each of the first 7 items has 2 possible responses (yes/no), while the 8th item is answered with a 5-point Likert scale. The possible total medication adherence score ranges between 0 and 8, and the higher the score, the better the adherence level. A total score < 6 is considered low adherence, while a total score of ≥ 6 but < 8 indicates moderate adherence, and a score of 8 indicates high adherence.
Time Frame: The outcome will be measured 1) following a month of polypill use, and 2) following a month of individual tablet use.
Population: Included participants who had this measure for both study periods (polypill and individual tablets).
Measure: Mean (95% Confidence Interval); unit: Total Score
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 26 | 26
Total Score | 4.1 [3.4 to 4.8] | 4.6 [3.9 to 5.4]

3. Secondary Outcome: Treatment Satisfaction Using the Treatment Satisfaction Questionnaire for Medication (TSQM 9)
Description: TSQM scores range from 0 to 100, with higher scores indicating greater treatment satisfaction.
Time Frame: The outcome will be measured 1) following a month of polypill use, and 2) following a month of individual tablet use.
Population: Included participants who had this measure for both study periods (polypill and individual tablets).
Measure: Mean (95% Confidence Interval); unit: Points on Global Satisfaction Score
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 26 | 26
Points on Global Satisfaction Score | 69.0 [61.6 to 76.3] | 73.6 [66.3 to 81]

4. Secondary Outcome: Heart Failure Admission Rate
Description: As a pilot trial, our study will not be powered for clinical outcomes, but key exploratory outcomes will include HFrEF admissions.
Time Frame: The outcome will be measured 1) following a month of polypill use, and 2) following a month of individual tablet use.
Population: For safety endpoints the number of participants included any participant who started that intervention period, so it is higher than then number analyzed who completed the efficacy outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 31 | 30
Participants | 0 | 1

5. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) 12
Description: Exploratory clinical outcomes will include change in health-related quality of life as measured by the Kansas City Cardiomyopathy Questionnaire. KCCQ scores range from 0 to 100, with higher scores indicating higher quality of life.
Time Frame: The outcome will be measured 1) following a month of polypill use, and 2) following a month of individual tablet use.
Population: Included participants who had this measure for both study periods (polypill and individual tablets).
Measure: Mean (95% Confidence Interval); unit: Overall Summary Score
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 26 | 26
Overall Summary Score | 67.9 [59.6 to 76.3] | 70.6 [62.2 to 78.9]

6. Secondary Outcome: Adherence Ratio to Individual Components of GDMT by Pill Count
Description: The investigators will calculate the adherence ratio for each individual component of GDMT (beta blocker, MRA, SGLT2i, and ACE/ARB/ARNI). This will be calculated as the (# pills missing) / (# pills supposed to be missing based on time elapsed between visits). This will allow us to investigate whether there is differential adherence to some categories of GDMT (for example, lower adherence to beta-blockers).
Time Frame: The outcome will be measured 1) following a month of polypill use, and 2) following a month of individual tablet use.
Population: Included participants who had this measure for both study periods (polypill and individual tablets); for beta blockers this is 23, ACE/ARB/ARNI 23, MRA 26, and SGLT2i 22.
Measure: Mean (95% Confidence Interval); unit: adherence ratio expressed in %
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 26 | 26
adherence ratio expressed in %
  Beta Blockers: number analyzed (Participants) | 23 | 23
  Beta Blockers | 73.8 [64.7 to 82.8] | 83.6 [74.6 to 92.7]
  ACE/ARB/ARNI: number analyzed (Participants) | 23 | 23
  ACE/ARB/ARNI | 71.1 [61.0 to 81.1] | 80.4 [70.4 to 90.4]
  MRA | 74.4 [66.3 to 82.5] | 83.7 [75.6 to 91.8]
  SGLT2i: number analyzed (Participants) | 22 | 22
  SGLT2i | 73.4 [64.5 to 82.3] | 81.6 [72.7 to 90.4]

7. Secondary Outcome: Blood Pressure (mmHg)
Description: Systolic Blood pressure at baseline and study follow-up
Time Frame: The outcome will be measured 1) following a month of polypill use, and 2) following a month of individual tablet use.
Population: Included participants who had this measure for both study periods (polypill and individual tablets).
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 26 | 26
mm Hg | 126 [118 to 134] | 124 [116 to 132]

8. Secondary Outcome: Heart Rate
Description: Heart rate (beats per minute)
Time Frame: The outcome will be measured 1) following a month of polypill use, and 2) following a month of individual tablet use.
Population: Included participants who had this measure for both study periods (polypill and individual tablets).
Measure: Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 25 | 25
beats per minute | 77 [71 to 84] | 77 [71 to 83]

9. Secondary Outcome: Weight
Description: Weight at baseline and study follow-up
Time Frame: The outcome will be measured 1) following a month of polypill use, and 2) following a month of individual tablet use.
Population: Included participants who had this measure for both study periods (polypill and individual tablets).
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 20 | 20
kg | 92.0 [82.8 to 101.1] | 93.0 [83.9 to 102.1]

10. Secondary Outcome: NT-ProBNP
Description: Lab test
Time Frame: The outcome will be measured 1) following a month of polypill use, and 2) following a month of individual tablet use.
Population: Included participants who had this measure for both study periods (polypill and individual tablets).
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 26 | 26
pg/ml | 1040.5 [448.4 to 1632.6] | 1086.5 [494.4 to 1678.7]

11. Secondary Outcome: Adverse Events
Description: The investigators will document adverse events throughout the study period, for example, hyperkalemia, dizziness, or other medication-related side effects. The investigators will ask participants about adverse events at in-person visits (0, 4, and 8 weeks) and at telephone calls at approximately 2 and 6 weeks.
Time Frame: 0, 2, 4, 6, and 8 weeks
Population: Safety endpoints include participants who started the intervention but did not complete it due to study dropout or loss to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 31 | 30
Participants
  Serious Adverse Events | 1 | 1
  Any Adverse Event | 6 | 7

12. Secondary Outcome: Total Daily Pill Burden of the Patient
Description: This will be calculated based on the patient's active medication list.
Time Frame: The outcome will be measured 1) following a month of polypill use, and 2) following a month of individual tablet use.
Population: Included participants who had this measure for both study periods (polypill and individual tablets).
Measure: Mean (95% Confidence Interval); unit: pills per day
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 27 | 27
pills per day | 10 [9 to 12] | 7 [5 to 8]

13. Secondary Outcome: Number of GDMT Pillars Prescribed
Description: The number of GDMT pillars prescribed to the patient (BB, MRA, SGLT2i, and either ACEi, ARB, or ARNI) will be calculated at baseline and week 4.
Time Frame: The outcome will be measured 1) at the start of the polypill intervention, and 2) at the start of the individual tablet intervention.
Population: This is measured at the start of each intervention period (because medication changes were only made for safety during each intervention period) so it includes all those who started each intervention period.
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 31 | 30
Participants
  Beta Blocker | 30 | 30
  ACE/ARB/ARNI | 28 | 28
  MRA | 30 | 29
  SGLT2i | 29 | 29

14. Secondary Outcome: HFrEF Polypill Patient Satisfaction Exit Survey
Description: A Likert scale-style exit survey will be administered asking participants to compare their experience with the HFrEF polypill vs. individual tablets. 4 questions will comprise an Acceptability of Intervention Measure (AIM): 1) the polypill met my approval; 2) the polypill was appealing to me; 3) I liked the polypill; and 4) I welcomed the polypill as a treatment option for my heart failure. Each question includes a 5-point Likert scale, from 1 (strongly disagree) to 5 (strongly agree). Participants' responses to the 4 AIM questions will be averaged to comprise an AIM summary score.
Time Frame: After study completion
Population: All participants who completed both intervention periods.
Measure: Median (Inter-Quartile Range); unit: Score on a 5-point scale
Groups:
- All Participants Who Completed the Study (Both Intervention Periods): All participants who completed the study for exit interviews/surveys
Arm/Group | All Participants Who Completed the Study (Both Intervention Periods)
Number analyzed (Participants) | 27
Score on a 5-point scale | 4.75 [4 to 5]

15. Secondary Outcome: Number of Participants Completing a Qualitative Exit Interview
Description: Participation in a semi-structured exit interview using a RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, Maintenance)
Time Frame: After study completion (between 8 and 12 weeks)
Population: All participants who completed both arms of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants Who Completed the Study (Both Intervention Periods)
Number analyzed (Participants) | 27
Participants | 27

16. Secondary Outcome: Implementation Outcome: Time Required to Manufacture the HFrEF Polypill at Our Community Pharmacy Partner
Description: Time required to prepare a 30-day supply of HFrEF polypill
Time Frame: Assessed at week 0 or week 4
Population: The pharmacy measured the time it took them to prepare the polypills for a subset of participants.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Manufacturing Set: The subset for which the pharmacy measured time to manufacture the polypills.
Arm/Group | Manufacturing Set
Number analyzed (Participants) | 9
minutes | 27 (4)

17. Secondary Outcome: Implementation Outcome: Cost of HFrEF Polypill Manufacturing at Our Community Pharmacy Partner
Description: Cost of manufacturing a 30-day supply of HFrEF polypill
Time Frame: Assessed at week 0 or week 4
Population: All participants who had polypills manufactured were included. The cost of manufacturing was the same for each patient, and was determined by the pharmacy partner (i.e. time and labor cost of preparing 1 month of polypill supply for 1 patient).
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Manufacturing Set
Number analyzed (Participants) | 30
Dollars | 60 (0)

18. Secondary Outcome: Number of Days Off of GDMT
Description: Number of days off GDMT due to a clinical event (e.g. hospitalization) or due to logistical / pharmacy issues
Time Frame: Assessed at weeks 4 and 8
Population: The analysis population includes all participants who started the intervention period and were not lost to follow up during that intervention period.
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Tablets | Polypill
Number analyzed (Participants) | 29 | 27
Participants
  0 days | 27 | 23
  1-3 days | 1 | 3
  4-7 days | 0 | 1
  8+days | 1 | 0

19. Other Pre Specified Outcome: Feasibility of Recruitment
Description: Number of months taken to recruit 30-40 people to consent to participate in the study
Time Frame: Completion of recruitment within 1 year of initiating recruitment
Population: This includes all participants who consented.
Measure: Number; unit: months
Groups:
- Consented: All participants who consented
Arm/Group | Consented
Number analyzed (Participants) | 35
months | 6

20. Other Pre Specified Outcome: Feasibility of Adherence to Study Protocols
Description: Successful completion of study related procedures for at least 20 participants (screening, randomization, drug allocation, follow-up procedures, retention, and transition to ongoing care)
Time Frame: Assessed following study completion (approximately 1 year)
Population: Number consented.
Measure: Count of Participants; unit: Participants
Arm/Group | Consented
Number analyzed (Participants) | 35
Participants | 27

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of starting the intervention period to the end of the intervention period.
Arm/Group | Individual Tablets | Polypill
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/31 | 1/30
Other Adverse Events (participants affected / at risk) | 5/31 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individual Tablets (N=31) | Polypill (N=30)
Heart Failure Hospitalization (Cardiac disorders) | 0 (0) | 1 (1)
Non-Heart Failure Hospitalization (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individual Tablets (N=31) | Polypill (N=30)
Non-HF Emergency Department or Urgent Care Visit (General disorders) | 1 (1) | 4 (4) — Assessed by asking participants and reviewing medical records
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 2 (2) — Acute Kidney Injury (serum creatinine increased >1.5x baseline
Hyperkalemia (Renal and urinary disorders) | 1 (1) | 1 (1) — Potassium > 5.5mEq/L
Dizziness or Hypotension (General disorders) | 2 (2) | 3 (3) — Dizziness or hypotension included patients who endorsed dizziness at a study visit or telephone follow-up, or were seen in the ER or urgent care for hypotension with BP < 90/60 (including during presentations for other diagnoses)
GDMT Medication Discontinuation or Downtriation due Intolerance (General disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
This study is a single-center, short-term pilot study in a safety-net setting with a meaningful dropout rate and high missingness of complete pill count data; blinding participants or investigators to the polypill vs individual tablets condition was not possible. Drug level monitoring was beyond the budget for this study. Finally, as a feasibility study, we included a number of secondary outcomes and did not correct for multiple comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT06029712/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT06029712/SAP_001.pdf
  • Informed Consent Form (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT06029712/ICF_002.pdf